CLINICAL TRIAL: NCT01739049
Title: The Influence of Appetite-Related Central and Gut Hormones in Modulating Binge Eating Behaviour in Obese and Overweight Healthy Subjects
Brief Title: Influence of Appetite Related Hormones in Binge Eating Behaviour Among the Overweight and Obese
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FF0192012
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Binge Eating Behaviour
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Liraglutide; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide and lifestyle counselling (Experimental): Liraglutide 0.6mg od for 1st week, then 1.2mg od for 2nd week then 1.8mg od until 12 weeks.
  Diet and Exercise
  Interventions: Drug: Liraglutide; Behavioral: Diet and Exercise
- Lifestyle counselling (Active Comparator): Diet and Exercise
  Interventions: Behavioral: Diet and Exercise

INTERVENTIONS:
Drug: Liraglutide — liraglutide
  Other Names: Victoza
  Arms: Liraglutide and lifestyle counselling
Behavioral: Diet and Exercise — diet and exercise

SUMMARY:
Malaysia has increasing challenges in lifestyle related diseases, which is related to eating habits and disorders. According to the National Health & Morbidity Survey in 2011; it was reported the prevalence of obesity is 15.1% in 2011; or 2.5 million of the population,; an increase of 7/9% when compared to the 14% prevalence in 2006. Binge eating is a symptom described in various eating disorders. It is an under-diagnosed medical condition closely linked to higher body mass index (BMI) or obesity as well as personality psychopathology, psychiatric and psychological disturbances. Meta-analysis has demonstrated that extremely strict restriction in dietary calorie and fat intake is needed to achieve meaningful weight loss. Appetite and satiety are influenced by extremely complex central and gut-related hormonal systems which modulate the regulation of food intake Centrally acting hormones include Neuropeptide Y (NPY), agouti gene-related peptide, orexin which are appetite-stimulating, melanocortins and alpha-melanocortin-stimulating hormone which promote satiety.

Gut-related peptides include ghrelin secreted by the stomach and the duodenum has orexigenic (appetite stimulating) effect; leptin secreted by adipose tissue has anorexic (appetite inhibiting) effect, cholecystokinin, glucagon-like peptide-1 (GLP-1) secreted by the proximal gastrointestinal tract which has slight anorexic effect, and peptide YY (PYY).

Appetite and obesity have also been commonly related to stress and may influence binge-eating episodes. Previous studies have demonstrated that high stress hormone cortisol is associated with increased appetite and cravings, with preference for high carbohydrate content, thus leading to weight gain.

In the previous study performed by our group on 738 normal subjects who were staffs of the Ministry of Health, Putrajaya, we found a prevalence of 19% binge eating behaviour, 83% of whom were either obese or overweight.

GLP-1 analogue used for the treatment of type 2 diabetes and is also shown to produce and maintain weight loss. Liraglutide, which provides a supra physiological amount of GLP-1 may cause appetite inhibition thus may benefit in reducing binge eating. The aim of this study is to closely observe the extensive profile of neuropeptide Y, ghrelin, leptin and GLP-1, influenced by a standard meal in binge eaters in comparison to non-binge eating controls. In addition, we aim to determine the association between binging and the respective appetite-related hormones and also cortisol. Finally we will also be assessing the efficacy of novel hormonal treatment of Liraglutide in reducing binge eating.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are willing to participate and sign informed consent form
* Subjects who are able to answer the questionnaire
* Subjects who are between 18-65 years old
* Subjects with BMI 30-45
* Subjects who are willing to administer injection

Exclusion Criteria:

* Pregnant subjects
* Subjects with chronic medical illness such as end stage renal failure, hepatic failure, diabetes mellitus, thyroidism, etc
* Subjects on medication that may influence appetite, satiety and weight
* Subjects that plan to move out of state/country

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Reduction in binge eating scale score | 12 weeks

SECONDARY OUTCOMES:
Reduction in weight | 12 weeks

OTHER OUTCOMES:
Profile of hormones | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nor Azmi Kamaruddin, Professor of Medicine, Principal Investigator — UKMMC; Rohana Abdul Ghani, Ass Professor of Medicine, Principal Investigator — UKMMC; Suehazlyn Zainuddin, MMed, Principal Investigator — UKMMC; Wan Nazaimoon Wan Mohamud, Phd Biochemistry, Principal Investigator — Institute for Medical Research, Inc.; Sarah Anne Robert, Mpharm, Principal Investigator — UKMMC
Locations (1):
- University Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robert SA, Rohana AG, Shah SA, Chinna K, Wan Mohamud WN, Kamaruddin NA. Improvement in binge eating in non-diabetic obese individuals after 3 months of treatment with liraglutide - A pilot study. Obes Res Clin Pract. 2015 May-Jun;9(3):301-4. doi: 10.1016/j.orcp.2015.03.005. Epub 2015 Apr 11. PMID 25870084